CLINICAL TRIAL: NCT04583215
Title: Enhancing Frontal Lobes Plasticity and Function in Patients With Mild Cognitive Impairment
Brief Title: Enhancing Frontal Lobes Plasticity in Mild Cognitive Impairment
Acronym: PAS-MCI
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Centre for Addiction and Mental Health (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: 050/2019
Record Dates: First submitted 2020-08-05; First posted 2020-10-12 (Actual); Last update posted 2024-10-26 (Actual); Status verified 2024-10

CONDITIONS: Mild Cognitive Impairment; Memory Impairment
Keywords: Memory Impairment; Executive Function; Transcranial Magnetic Stimulation; Paired Associative Stimulation; Neuroplasticity; Electroencephalography; Working Memory; Cognition; Prefrontal Cortex
MeSH Terms: conditions — Cognitive Dysfunction; Memory Disorders | interventions — Transcranial Magnetic Stimulation

STUDY DESIGN:
Intervention Model Description: At screening 100 MCI and 50 HC participants will undergo clinical and cognitive assessments and a brain MRI to localize the DLPFC. If eligible, at baseline, all participants will undergo N-back and PAS-EEG to assess baseline DLPFC plasticity. Following baseline procedures, MCI participants will be randomized (1:1) to the study intervention consisting of 10 sessions of either bilateral PAS or PAS-C to the right and left DLPFC, 1 session/day, for 10 days. On the last day of the intervention, participants will repeat the cognitive assessments and on the following day they will repeat N-back and PAS-EEG to assess the effect of daily PAS on executive function and DLPFC plasticity. Finally, on the 7th day following the intervention (Visit 16), MCI participants will repeat N-back and PAS-EEG, and on the 28th and 29th day (Visit 17 and Visit 18) following the intervention, MCI participants will repeat the cognitive assessments, N-back and PAS-EEG to evaluate the sustainability of effects.
Who Masked: Participant, Investigator, Outcomes Assessor
Masking Description: A unique advantage of Paired Associative Stimulation (PAS) over other TMS-based interventions is that its control condition (PAS-C) is almost impossible to distinguish from active PAS. Thus, the RCT phase of the study will be completed under triple-blind conditions. First, participants will be blind to whether they are randomized to PAS or PAS-C. Second, the investigator team (investigators and interventionists delivering the 10-session course) will be blind to group assignment. Third, the outcomes assessors conducting the clinical, cognitive and PAS-EEG assessments at baseline and follow-ups will be blind to group assignment.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (3):
- Active PAS (Active Comparator): After completing the N-back and PAS-EEG at Visit 4, MCI participants randomized to the active condition will receive a 10-session course of PAS (Visits 5-14), followed by the three follow-up assessments at 0 days, 7 days, and 28 days post intervention.
  Interventions: Device: Paired Associative Stimulation (PAS)
- PAS-Control (PAS-C) (Sham Comparator): After completing the N-back and PAS-EEG at Visit 4, MCI participants randomized to the sham condition will receive a 10-session course of PAS-C (Visits 5-14), followed by the three follow-up assessments at 0 days, 7 days, and 28 days post intervention.
  Interventions: Device: Paired Associative Stimulation (PAS)
- Healthy Control (No Intervention): Healthy Controls will complete screening and baseline N-Back and PAS-EEG. 10 HC participants will also complete the optional pilot eye tracking VPC assessment following N-Back at the Baseline visit. HC participants will not complete the 10-session course of PAS or follow-up assessments.

INTERVENTIONS:
Device: Paired Associative Stimulation (PAS) — On each of the 10 days of the intervention, participants will receive PAS (or PAS-C) to the left DLPFC by delivering peripheral nerve stimulation (PNS) to the right median nerve and TMS to the left DLPFC, followed immediately by PAS (or PAS-C) to the right DLPFC by delivering PNS to the left median nerve and TMS to the right DLPFC. PAS-C differs from PAS only by including an interstimulus interval of 100 ms between PNS and TMS to the DLPFC, compared to 25 ms in the active PAS condition. Using 100 ms interval, we have previously demonstrated that PAS-C does not induce PAS-LTP in the DLPFC. If a participant cannot attend one or more of the 10 consecutive PAS or PAS-C treatment sessions, we will allow up to four extra treatment days to make up for missed sessions.
  Other Names: Transcranial Magnetic Stimulation (TMS); Peripheral Nerve Stimulation (PNS)
  Arms: Active PAS; PAS-Control (PAS-C)

SUMMARY:
More than 5 million people live with Alzheimer's dementia (AD) in North America. No effective treatment exists yet probably because by the time AD has developed it is too late to intervene. Mild Cognitive Impairment (MCI) is a clinical state that typically precedes AD. In MCI, the prefrontal cortex supports compensatory mechanisms that depend on robust synaptic plasticity and that delay progression to AD. Using a neurostimulation approach that enhances prefrontal cortical plasticity in vivo, this project aims to enhance prefrontal cortical plasticity and function in patients with MCI. If successful, this project would discover a treatment modality that enhances compensation in MCI and ultimately, prevents progression to AD.

DETAILED DESCRIPTION:
Paired Associative Stimulation (PAS) is a neurostimulation approach that induces cortical plasticity by simulating spike-timing-dependent plasticity. Combining PAS with electroencephalography (EEG) (PAS-EEG), we can assess dorsolateral prefrontal cortex (DLPFC) plasticity in vivo. Using PAS-EEG, we have demonstrated that patients with AD are impaired on DLPFC plasticity compared to healthy control (HC) individuals and that DLPFC plasticity is associated with working memory in AD and HC individuals. We have also shown that a 2-week course of daily PAS to the left DLPFC restores DLPFC plasticity in patients with AD and enhances their working memory.

Thus, we propose to study DLPFC plasticity and its relationship to executive function in MCI and then assess the efficacy of a 2-week course of PAS in enhancing DLPFC plasticity and executive function in this population.

If successful, this project will identify a novel neurostimulation intervention (PAS) to enhance prefrontal cortical function in MCI patients. This enhancement could result in modifying the trajectory of Alzheimer's disease by delaying the progression from MCI to clinical AD. This project will also identify a mechanism (neuroplasticity) that underlies enhanced prefrontal cortical function. Other interventions (e.g. behavioral, neurostimulation, pharmacological) could then be tested whether they engage neuroplasticity to enhance prefrontal cortical function.

The primary objectives and hypotheses of the study are as follows:

Objective 1: To compare baseline DLPFC plasticity and its relationship to executive function in MCI vs. HC participants. Hypothesis 1a: MCI participants will be impaired on PAS-LTP (TMS-induced cortical evoked activity) in the left DLPFC compared to HC participants. Hypothesis 1b: MCI participants will be impaired on 2-back d' compared to HC participants. Hypothesis 1c: MCI participants will be impaired on a composite executive function measure compared to HC participants. Hypothesis 1d: PAS-LTP will be associated with 2-back d' in MCI and HC participants after controlling for age, sex, and education. Hypothesis 1e: PAS-LTP will be associated with composite executive function measure in MCI and HC participants after controlling for age, sex, and education.

Objective 2: To assess the efficacy of a 10-session course of bilateral PAS in enhancing DLPFC plasticity and executive function in MCI participants. Hypothesis 2a: MCI participants randomized to 10-session course of active PAS will experience higher PAS-LTP in the left DLPFC immediately and 1 and 4 weeks after the course compared to MCI participants randomized to a 10-session course of PAS-C. Hypothesis 2b: MCI participants randomized to a 10-session course of active PAS will experience better 2-back performance immediately and 1 and 4 weeks following the 10-session course compared to MCI participants randomized to the course of PAS-C. Hypothesis 2c: MCI participants randomized to a 10-session course of active PAS will experience higher composite executive function scores immediately and 1 and 4 weeks following the 10-session course compared to MCI participants randomized to the course of PAS-C.

Objective 3: To assess whether changes in DLPFC plasticity mediate changes in executive function in MCI participants following the 10-session course. Hypothesis 3a: Changes in PAS-LTP immediately and 1 and 4 weeks following the 10-session course will mediate changes in 2-back d' at all of these three follow-up time points. Hypothesis 3b: Changes in PAS-LTP immediately and 1 and 4 weeks following the 10-session course will mediate changes in composite executive function measure at all of these three follow-up time points. Conditions/focus of study (primary disease or condition being studied).

Objective 4: Evaluating eye movement in addition to EEG as a potential cognitive biomarker in unimpaired versus MCI older adults using the visual paired comparison (VPC) eye tracking task. As a powerful eye tracking approach, the VPC (commonly referred to as the preferential viewing task) is a nonverbal recognition task that has demonstrated promising evidence for detecting cognitive impairments associated with MCI through analyzing eye movement patterns. Hypothesis 4a: Older individuals with MCI will exhibit diminished eye movement markers (diminished preference for viewing novel versus familiarized stimuli) and EEG markers (P300 and synchrony of theta oscillations) of memory compared to healthy individuals. Hypothesis 4b: Preferential viewing for novel stimuli will be positively associated with EEG markers of memory (P300 and synchrony of theta oscillations). The eye tracking VPC task will first be piloted in older healthy controls in order to optimize the parameters of the eye tracking technology to ensure optimal performance prior to administering in MCI individuals.

Exploratory Objective 5: 5a: We will explore, in both HC and MCI participants, the relationships between wisdom as measured using the Jeste-Thomas Wisdom Index (JTWI) before baseline PAS-EEG and DLPFC plasticity at baseline. 5b: We will explore, in both HC and MCI participants, change in wisdom on JTWI as administered after baseline PAS-EEG in response to single PAS session. 5c: We will explore, in MCI participants only, change in wisdom after the 10-session course of PAS or PAS-C by administering JTWI before and after each follow-up PAS-EEG session.

ELIGIBILITY:
MCI Group:

Inclusion Criteria:

1. Age 60 years or above.
2. Right-handed (to minimize heterogeneity with respect to cognitive reserve and plasticity) and as determined by the Edinburgh Handedness Questionnaire.
3. Diagnosis of MCI due to AD using the core clinical criteria by the National Institute on Aging and Alzheimer's Association for MCI participants (NIA-AA) and ascertained by a study investigator. The following checklist will be used to ascertain the MCI diagnosis:

   1. Cognitive concern reflecting a change in cognition reported by patient or informant or clinician (i.e., historical or observed evidence of decline over time).
   2. Not demented ascertained using the study investigator opinion.
   3. No vascular, traumatic, or medical causes of cognitive decline ascertained using the study investigator opinion.
   4. Evidence of longitudinal decline in cognition, when feasible, and ascertained using the study investigator opinion.
4. Objective evidence of single or multi domain MCI, where single domain MCI refers to deficits using NP battery on only one of the cognitive domains (Speed of Processing; Working Memory; Executive Functioning; Verbal Memory; Visual Memory; Language)and multi domain MCI refers to deficits in more than one of these domains. To determine impairment in one or more cognitive domain, after the NP battery is administered and double scored, a consensus meeting will be held with the research study staff, the study Principal Investigator and the study Neuropsychologist during which eligibility will be discussed. The meeting attendees will take into consideration the participant's education, parental education, pre-morbid IQ, physician's assessment and NP scores to determine if the participant has impairment in one or more cognitive domain.
5. Willingness to provide informed consent.
6. Ability to read and communicate in English (with corrected vision and hearing, if needed).

Exclusion Criteria:

1. Current use of an acetylcholine esterase inhibitor or memantine ascertained using a Medication List.
2. Major Depressive Disorder with active symptoms in the last 3 months ascertained using the Structured Clinical Interview for DSM 5 (SCID-5).
3. A lifetime diagnosis of bipolar disorder; intellectual disability; or a psychotic disorder ascertained using the SCID-5.
4. Substance use disorder active in the last 3 months ascertained using the SCID-5.
5. Any other DSM-5 diagnosis ascertained using the SCID-5 that may be associated with prefrontal cortical dysfunction as ascertained using a study investigator opinion.
6. Current anticonvulsant use due to its impact on TMS induced activity and ascertained using a Medication List. An exception will be made if they are taking gabapentin or pregabalin AND if the dose had been stable for at least 4 weeks prior to study entry AND if prescribed for chronic pain.
7. Current benzodiazepine use of more than what is equivalent to lorazepam 2 mg/day as ascertained using a Medication List. This is due to their known pro-GABAergic activity and the suppressive effect of GABAergic agents on cortical plasticity.
8. Any contraindication to MRI or contraindication to TMS (e.g., cardiac pacemaker, acoustic device, history of seizures) ascertained using the TMS Adult Safety Screen (TASS).

Healthy Controls

Inclusion Criteria:

1. Age 60 years or above.
2. Right-handed (to minimize heterogeneity with respect to cognitive reserve and plasticity) and as determined by the Edinburgh Handedness Inventory.
3. MoCA score > 26.
4. Ability to read and communicate in English (with corrected vision and hearing, if needed).
5. Willingness to provide informed consent.

Exclusion Criteria:

1. Diagnosis of MCI due to AD using the core clinical criteria by the National Institute on Aging and Alzheimer's Association for MCI participants and ascertained by a study investigator.
2. Any lifetime DSM-5 diagnosis ascertained using the SCID-5 (except for simple/specific phobias) or diagnosis that may be associated with prefrontal cortical dysfunction as ascertained using a study investigator opinion.
3. Any current use of a psychotropic medication for a CNS condition as ascertained using the Medication List.
4. Current anticonvulsant use due to its impact on TMS induced activity and ascertained using a Medication List. An exception will be made if they are taking gabapentin or pregabalin AND if the dose had been stable for at least 4 weeks prior to study entry AND if prescribed for chronic pain.
5. Current benzodiazepine use of more than what is equivalent to lorazepam 2 mg/day as ascertained using a Medication List. This is due to their known pro-GABAergic activity and the suppressive effect of GABAergic agents on cortical plasticity.
6. Any contraindication to MRI or contraindication to TMS (e.g., cardiac pacemaker, acoustic device, history of seizures) ascertained using the TMS Adult Safety Screen (TASS).

Min Age: 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 150 (Estimated)
Dates: Start 2020-10-12 (Actual); Primary Completion 2026-10-01 (Estimated); Study Completion 2026-12-01 (Estimated)

PRIMARY OUTCOMES:
PAS-Long-term-potentiation (PAS-LTP) | Baseline
  PAS-LTP is measured as the ratio of TMS-induced cortical evoked activity (CEA) post-PAS to TMS-induced CEA pre-PAS
Change in PAS-Long-term-potentiation (PAS-LTP) | Baseline, immediately and 1 and 4 weeks following the 10-session course
  PAS-LTP is measured as the ratio of TMS-induced cortical evoked activity (CEA) post-PAS to TMS-induced CEA pre-PAS
N-Back Performance | Baseline
  The primary outcome measure will be based on the 2-back condition of the N-Back. N-back accuracy will be assessed using d', which is a sensitivity index based on the z scores of hit rates (H- correctly responding to target trials as target trials) and false alarm rates (F- incorrectly responding to non-target trials as target trials) using the following formula: d' = z(H) - z(F).
Change in N-Back Performance | Baseline, immediately and 1 and 4 weeks following the 10-session course
  The primary outcome measure will be based on the 2-back condition of the N-Back. N-back accuracy will be assessed using d', which is a sensitivity index based on the z scores of hit rates (H- correctly responding to target trials as target trials) and false alarm rates (F- incorrectly responding to non-target trials as target trials) using the following formula: d' = z(H) - z(F).

SECONDARY OUTCOMES:
Executive Function Composite Measure | Baseline
  The executive function composite measure will be calculated using established and well validated tests from a comprehensive neuropsychological battery.
Change in Executive Function Composite Measure | Baseline, immediately and 4 weeks following the 10-session course
  The executive function composite measure will be calculated using established and well validated tests from a comprehensive neuropsychological battery.

CONTACTS AND LOCATIONS:
Overall Officials: Sanjeev Kumar, MD, Principal Investigator — Centre for Addiction and Mental Health
Locations (1):
- Centre for Addiction and Mental Health, Toronto, Ontario, Canada

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Rajji TK, Sun Y, Zomorrodi-Moghaddam R, Farzan F, Blumberger DM, Mulsant BH, Fitzgerald PB, Daskalakis ZJ. PAS-induced potentiation of cortical-evoked activity in the dorsolateral prefrontal cortex. Neuropsychopharmacology. 2013 Nov;38(12):2545-52. doi: 10.1038/npp.2013.161. Epub 2013 Jul 3. PMID 23820586
- [Background] Kumar S, Zomorrodi R, Ghazala Z, Goodman MS, Blumberger DM, Cheam A, Fischer C, Daskalakis ZJ, Mulsant BH, Pollock BG, Rajji TK. Extent of Dorsolateral Prefrontal Cortex Plasticity and Its Association With Working Memory in Patients With Alzheimer Disease. JAMA Psychiatry. 2017 Dec 1;74(12):1266-1274. doi: 10.1001/jamapsychiatry.2017.3292. PMID 29071355